CLINICAL TRIAL: NCT04523272
Title: A Randomized, Positive Parallel Controlled, Multicenter Phase III Study of TQB2450 Injection Combined With Anlotinib Hydrochloride Capsule Versus Sunitinib in Subjects With Advanced Renal Cancer
Brief Title: A Study of TQB2450 Injection Combined With Anlotinib Hydrochloride Capsule Versus Sunitinib in Subjects With Advanced Renal Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TQB2450-III-07
Record Dates: First submitted 2020-08-20; First posted 2020-08-21 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Advanced Renal Cancer
MeSH Terms: interventions — anlotinib; Sunitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQB2450 + Anlotinib (Experimental): TQB2450 1200 mg administered intravenously (IV) on Day 1 of each 21-day cycle ,Anlotinib capsules 12 mg given orally, once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21).
  Interventions: Drug: TQB2450; Drug: Anlotinib
- Sunitinib Malate Capsules (Active Comparator): Sunitinib malate capsule 50mg administered orally, once daily in 28-day cycle(14 days on treatment from Day 1-14, 14 days off treatment from day 15-28).
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: TQB2450 — TQB2450 is a humanized monoclonal antibody targeting programmed death ligand-1 (PD-L1), which prevents PD-L1 from binding to PD-1 and B7.1 receptors on T cell surface, restores T cell activity, thus enhancing immune response and has potential to treat various types of tumors.
  Arms: TQB2450 + Anlotinib
Drug: Anlotinib — A multi-target receptor tyrosine kinase inhibitor.
  Arms: TQB2450 + Anlotinib
Drug: Sunitinib — A multi-target receptor tyrosine kinase inhibitor.
  Arms: Sunitinib Malate Capsules

SUMMARY:
This study is a randomized, positive parallel controlled, multicentre phase III clinical trial to evaluate the efficacy and safety of TQB2450 combined with anlotinib versus sunitinib in subjects with advanced renal cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. Histopathologically confirmed renal clear cell cancer, including advanced renal cell carcinoma with clear cell components.

  2. Has not receiving systemic therapy for local advanced/metastatic disease. 3. At least has one measurable lesion. 4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1; Life expectancy ≥ 3 months.

  5. Adequate laboratory indicators. 6. Agree to provide at least 5 slices tumor tissue samples for biomarker detection.

  7. Serum or urine pregnancy tests are negative within 7 days before randomization; Men and women should agree to use effective contraception during the study period and after the end of the study period within 6 months.

  8. Understood and signed an informed consent form.

Exclusion Criteria:

* 1. Has symptomatic central nervous system (CNS) disease and / or cancerous meningitis, pia mater disease.

  2. Has received anti-angiogenesis targeted therapy or targeted PD-1 and PD-L1 immunotherapy.

  3. Has active virus, bacteria, fungal infection; Cardiovascular and cerebrovascular diseases; Gastrointestinal abnormalities; Immunodeficiency; Bleeding risk; Lung disease; Neurological or psychiatric disorders.

  4. Has participated in other clinical trials within 30 days before randomization.

  5. Has received attenuated live vaccine within 28 days before randomization or planned to received attenuated live vaccine during the study period.

  6. Pregnant or lactating women. 7. According to the judgement of the investigators, there are other factors that may lead to the termination of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 528 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) evaluated by Independent Review Committee(IRC) | up to 60 weeks
  PFS defined as the time from randomization until the first documented progressive disease (PD) or death from any cause, based on IRC.

SECONDARY OUTCOMES:
Progression free survival (PFS) evaluated by investigator | up to 60 weeks
  PFS defined as the time from randomization until the first documented progressive disease (PD) or death from any cause, based on investigator.
Overall survival (OS) | up to 60 weeks
  OS defined as the time from randomization to death from any cause. Participants who do not die at the end of the extended follow-up period, or were lost to follow-up during the study, were censored at the last date they were known to be alive.
Disease control rate（DCR） | up to 60 weeks
  Percentage of participants achieving complete response (CR) and partial response (PR) and stable disease (SD).
Duration of response（DOR） | up to 60 weeks
  The time when the participants first achieved complete or partial remission to disease progression.
Progression-free survival at 12 months | up to 12 months
  Percentage of participants whose PFS has achieved at least 12 months.
Overall survival at 12 months | up to 12 months
  Percentage of participants whose OS has achieved at least 12 months.
Overall survival at 24 months | up to 24 months
  Percentage of participants whose OS has achieved at least 24 months.

CONTACTS AND LOCATIONS:
Locations (39):
- China (39):
  - The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of the Chinese People's Liberation Army Army Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - First Hospital of Lanzhou University, Lanzhou, Gansu
  - Sun Yat-sen of Cancer Center, Guangzhou, Guangdong
  - The Affiliated Tumor Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Tenth People's Hospital of Tongji University, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital of Xi 'an Jiaotong University, Xi’an, Shanxi
  - The First Affiliated Hospital of PLA Air Force Military Medical University, Xi’an, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Second Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - First Affiliated Hospital,School of Medicine,Shihezi University, Shihezi, Xinjiang
  - The Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Cancer Hospital of The University of Chinese Academy of Sciences, Hangzhou, Zhejiang
  - The First Hospital of Jiaxing, Jiaxing, Zhejiang

REFERENCES:
- [Derived] Zhou A, Shen P, Li J, Qu W, Wang Z, Ren X, Li Y, Jiang S, Li G, Zeng Y, Qin W, Wu J, Chen P, Zhou F, Guo H, Ji Z, Wang Y, He Z, Wu J, Shi B, Liu L, Yao X, Ma L, Liu Z, Gou X, Fu B, Wang S, Jiang K, Chong T, Tu X, Zhang X, Yu D, Rexiati M, Xue X, Fei J, Wan J, Jia L, He Y, Cui T, Yang AQ, Guo J, Sheng X. First-line benmelstobart plus anlotinib versus sunitinib in advanced renal cell carcinoma (ETER100): a multicentre, randomised, open-label, phase 3 trial. Lancet Oncol. 2025 Sep;26(9):1145-1157. doi: 10.1016/S1470-2045(25)00343-2. PMID 40907513